CLINICAL TRIAL: NCT02902861
Title: An International Prospective, Double-blind, Placebo-controlled Phase III Randomised Controlled Trial (RCT) in Patients With Moderate to Severe Psoriasis Are Treated With Subcutaneous (s.c.) Methotrexate Using an Optimized Treatment Schedule.
Brief Title: Trial in Patients With Psoriasis Treated With Methotrexate Using an Optimized Treatment Schedule (METOP)
Acronym: METOP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prof. Kristian Reich (Industry)
Responsible Party: Sponsor-Investigator, Prof. Kristian Reich, Professor, Sciderm GmbH
Organization: Sciderm GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 165-001; 2012-002716-10 (EudraCT Number)
Record Dates: First submitted 2016-07-26; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- methotrexate (Active Comparator): Once weekly (every 7 days) s.c. administration of 17.5 mg MTX. If PASI50 is not reached after 8 weeks (week 8) or PASI75 is not reached after 24 weeks, the dosing will be increased to 22.5 mg MTX/week. If patients were already dosed with 22.5 mg MTX/week in week 24 and PASI50 is not reached, patients will be excluded from treatment. Primary endpoint after 16 weeks.
  Interventions: Drug: Methotrexate
- Placebo (NaCl-Solution) (Placebo Comparator): Once weekly (every 7 days) s.c. administration of 0.35 mL placebo If PASI50 is not reached after 8 weeks (week 8), the dosing will be increased to 0.45 mL placebo/week. Primary endpoint after 16 weeks. After 16 weeks patients will receive 17.5 mg MTX / week. If PASI50 is not reached after 8 weeks of MTX treatment (week 24), uptitration to 22.5 mg MTX/ 0.45 mL Plac / week will be done. Patients, who will reach PASI75 under placebo treatment after 16 weeks, will be dosed neither with placebo nor with MTX until relapse. After relapse the patients will be dosed with a starting dose of 17.5 mg MTX / week.
  Interventions: Drug: Placebo ( for Methotrexate)

INTERVENTIONS:
Drug: Methotrexate — methotrexate 50 mg/ml in syringes for sub-cutaneous injection; Once weekly (every 7 days) s.c. administration of 17.5 mg MTX; If PASI50 is not reached after 8 weeks, the dosing will be increased to 22.5 mg
  Other Names: MTX
  Arms: methotrexate
Drug: Placebo ( for Methotrexate) — NaCl-Solution manufactured to mimic Methotrexate
  Arms: Placebo (NaCl-Solution)

SUMMARY:
This is a multicenter, multinational (12 centers planned, in Germany 9 centers and in France, the Netherlands and the United Kingdom (UK) 1 center in each country respectively), randomized, double-blinded, placebo-controlled study. The primary objective is to evaluate the efficacy of methotrexate (MTX) in patients with moderate to severe Psoriasis compared to Placebo as assessed by the primary endpoint "75% reduction of Psoriasis Area Severity Index" (PASI 75 ) during a 16 week treatment phase. As secondary objectives the safety and efficacy of the optimized treatment schedule will be assessed using multiple methods (e.g. (Serious) Adverse Events ((S)AE) occurrence and questionnaires)

DETAILED DESCRIPTION:
The present study was initiated to further increase the knowledge about the optimal dosing regimen and to thus optimize the efficacy and safety of MTX treatment for patients with moderate to severe psoriasis. In view of the described risk-benefit profile of MTX, an initial dose of at least 15 mg per week administered subcutaneously followed by 5 mg folic acid p.o. 24 hours after MTX application seems appropriate. Since 20 mg MTX per week has been proven to be beneficial in a considerable part of patients, who did not respond sufficiently to 15 mg MTX per week, in this study the dosing starts with a dose of 17.5 mg MTX per week, administered subcutaneously. At such a starting dose, it was expected to find the highest MTX efficacy possible, but with appropriate safety margins. If in a patient, a "50% reduction of Psoriasis Area Severity Index" PASI50 response is not achieved in week 8, the dose will be increased to 22.5 mg MTX per week. All dosages used in this study lay within the approved dosing range of MTX. The study will be conducted in a double-blind, placebo controlled manner. Placebo was chosen as control since only this comparator allows a reliable interpretation of safety and efficacy data.

ELIGIBILITY:
Inclusion Criteria:

1. Are 18 years of age or older at time of informed consent; may be men or women.
2. Are MTX naïve
3. Moderate to severe plaques psoriasis (according rule of ten (PASI ≥10 or BSA ≥ 10 or DLQI ≥ 10) for at least 6 months with or without psoriatic arthritis (however, highly active psoriatic arthritis is excluded, defined by. > 5 swollen tender joints or soles and C-Reactive Protein (CRP) >2 x UNL) .
4. Women of childbearing potential and all men must be using a highly effective method of contraception (pearl index < 1%) as defined blow and must agree to continue to use such measures and not become pregnant or plan a pregnancy until 6 months after receiving the last injection of Investigational Medicinal Product (IMP).Highly effective method is defined as: Use of oral, injected or implanted hormonal methods, intrauterine device (IUD) or intrauterine system (IUS), barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
5. Able to adhere to the study visit schedule and other protocol requirements.
6. Capable of giving informed consent. The informed consent must be obtained prior to any study related procedures.
7. Must avoid prolonged sun exposure and avoid use of tanning booths or other ultraviolet light sources during study.
8. Must agree not to receive a live virus or live bacterial vaccination 4 weeks prior to the first IMP s.c. administration, during the trial and up to 3 months after the last injection.
9. Chest X-ray investigation within the last 6 months prior to first s.c. administration of IMP and show no clinically relevant abnormalities

Exclusion Criteria:

1. Currently have non-plaque forms of psoriasis (eg, erythrodermic, guttate, or pustular).
2. Have current drug-induced psoriasis (eg, a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, (hydroxy-) chloroquine, or lithium).
3. Are pregnant, nursing, or planning pregnancy (both men and women) while enrolled in the study.
4. Have screening laboratory test results for the following parameters outside the stated ranges (please refer also to :

   1. Hemoglobin < 10 g/dL
   2. White blood cells < 3.0 x 109/L
   3. Neutrophils < 1.5 x 109/L
   4. Platelets < 100 x 109/L
   5. Creatinine clearance (calculated according to Cockcroft-Gault) < 50 mL/min)
   6. Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), and Gamma Glutamyltransferase (γ-GT) levels must be > 2 times the upper limit of normal range
   7. Bilirubin > 5mg/dl (85,5 μmol/l)
   8. Hypalbuminemia <3,5 g/dl
5. Have used any other IMP within the previous 4 weeks or 5 times the half-life of an investigational agent prior to the first s.c. administration of the IMP of this study, whichever is longer.
6. Not able or willing to wash out any prohibited medications as listed below.

   * Any biologics; washout 5 times of half-life
   * Phototherapy or any systemic medications that could affect the psoriasis (including but not limited to oral or injectable corticosteroids, retinoids, 1,25 dihydroxy vitamin D3 and analogues, sulfasalazine, hydroxyurea, or fumaric acid derivates), within 4 weeks
   * Any topical medications that could affect the psoriasis (e.g. corticosteroids, anthralin, calcipotriene, topical vitamin D derivates, retinoids, tazarotene), within 2 weeks
   * Any systemic immunosuppressants (e.g. azathioprine, cyclosporine, 6-thioguanine, mercaptopurine, mycophenolate mofetil, hydroxyurea, and tacrolimus) ,within 4 weeks
   * lithium, antimalarial agents To be stopped directly prior to first s.c. administration of IMP
   * Intramuscular gold ,Within 4 weeks Patients who take prohibited medications that cannot be washed out within 4 weeks or at least 5 times of the half-life of the investigational agent prior to first s.c.

   administration of IMP should not be asked to participate in the trial.
7. Have a history of chronic or recurrent infectious disease or had a serious infection or have been hospitalized or received i.v. antibiotics for the treatment of an infection within 2 months prior to screening.
8. History of radiotherapy or planed concomitant radiotherapy
9. Ulcers of the oral cavity (e.g. ulcerative stomatitis) and/or known gastrointestinal ulcer disease
10. A known B12/cobalamin deficiency
11. Known diagnosed ascites or pleural effusions
12. Have a history of latent or active Tuberculosis (TB) (prior to screening).
13. Have current signs or symptoms of severe, progressive, or uncontrolled renal (specifically with calculated creatinine clearance < 20), hepatic (especially with bilirubin > 5mg/dl (85,5 mol/l), hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease.
14. Have any known malignancy or have a history of malignancy (with the exception of basal cell carcinoma, squamous cell carcinoma in situ of the skin, or cervical carcinoma in situ that has been treated with no evidence of recurrence, or squamous cell carcinoma of the skin that has been treated with no evidence of recurrence within 5 years prior to the first administration of study agent).
15. Have shown a previous immediate hypersensitivity response, including anaphylaxis, to the folic acid
16. Are unable or unwilling to undergo multiple venipunctures because of poor tolerability or lack of easy access to veins.
17. Are known to have had a substance abuse (drug or alcohol) problem within the previous 12 months.
18. Staff or relatives/partner of any clinical research site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Difference in 75% reduction of Psoriasis Area Severity Index (PASI75) responder rate between treatment arms | week 16

SECONDARY OUTCOMES:
Difference in PASI75 responder rate between treatment arms | weeks 52
Difference in 50% reduction of Psoriasis Area Severity Index (PASI50) | weeks 15 and 52
Difference in 90% reduction of Psoriasis Area Severity Index (PASI90) | weeks 15 and 52
PASI75 in placebo arm (cross-over) | weeks 32
Difference in Nail Psoriasis Severity Index (NAPSI) | weeks 16 and 52
Difference in Body Surface Area Index (BSA) | weeks 16 and 52
Difference in Physician's Global Assessment (PGA) | weeks 16 and 52
Difference in Psoriatic Arthritis Index (PsA) | weeks 16 and 52
Difference in Patient's satisfaction with metex® pre-filled syringe (PSAT metex®) | weeks 16 and 52
Difference in Dermatology Life Quality Index (DLQI) | weeks 16 and 52
Difference in European Qualification-5D-Questionnaire (EQ-5D) | weeks 16 and 52
Safety and tolerability assessed by Adverse Events (AE)/ Serious Adverse Events (SAE) tolerability at the site of administration | week 0 - week 51
Safety and tolerability assessed by laboratory values | week 0 - week 51
local tolerability at the site of administration assessed by Erythema | week 0 - week 51
  Erythema (redness): diameter (mm) and severity from none to severe (0 = none,
  1= mild, 2 = moderate 3 = severe)
local tolerability at the site of administration assessed by Swelling | week 0 - week 51
  Swelling/Induration: diameter (mm) and severity from none to severe (0 = none,
  1= mild, 2 = moderate 3 = severe)
local tolerability at the site of administration assessed by Hematoma | week 0 - week 51
  Hematoma: yes/ no and if present diameter (mm)
local tolerability at the site of administration assessed by Local Pain | week 0 - week 51
  Local pain - assessed by the study subject on a visual analogue scale (1-10)
local tolerability at the site of administration assessed by Pruritus | week 0 - week 51
  Pruritus - assessed by the study subject on a visual analogue scale (1-10)
Changes of levels of molecular biologic analysis | at baseline and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Mrowietz, Professor, Principal Investigator — Psoriasis-Zentrum, Universitäts-Hautklinik Kiel
Locations (1):
- Psoriasis-Zentrum, Universitäts-Hautklinik Kiel, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No